CLINICAL TRIAL: NCT00758030
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Dose Study to Evaluate and Compare the Pharmacokinetics of ER OROS Paliperidone in Healthy Japanese and Caucasian Subjects.
Brief Title: Study Evaluating and Comparing Single Dose and Multiple Dose Pharmacokinetics of ER OROS Paliperidone in Healthy Japanese and Caucasian Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004933
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: Paliperidone ER OROS

SUMMARY:
The purpose of the study was to evaluate and compare the pharmacokinetics of ER OROS paliperidone in healthy Japanese and Caucasian patients.

DETAILED DESCRIPTION:
This was a randomized (study medication assigned by chance), double blind (neither physician or patient knows the name of the study medication/placebo assigned) study comparing the single does (SD) and multiple dose (MD) pharmacokinetics of ER OROS paliperidone in 30 healthy Japanese and 30 healthy Caucasian adults.. The primary objectives of this study were to 1) evaluate the safety and tolerability of extended-release (ER) OROS paliperidone in healthy Japanese adults, 2) to evaluate the single dose (SD) and multiple dose (MD) pharmacokinetics of ER OROS paliperidone in healthy Japanese adults, and 3) to compare the SD and MD pharmacokinetics of ER OROS paliperidone in healthy Japanese and Caucasian adults. Of the 30 Japanese patients enrolled, at least 10 were to be men and 10 to be were women. An equal number of Caucasian patients, matched as closely as possible to the Japanese subjects for sex, age, and weight, were enrolled. Patients were randomly assigned to receive either ER OROS paliperidone or placebo (4:1 ratio). Blood samples for the determination of paliperidone enantiomer plasma concentrations were collected immediately prior to dosing on Days 1, 9, 10, 11, and 19, and at 2, 4, 6, 9, 12, 16, 18, 20, 22, 24, 27, 33, 36, 48, 58, 72, and 96 hours after dosing on Days 1, 11, and 19. Urine samples were collected predose and over 0-12, 12-24, 24-36, and 36-48 hour intervals after dosing on Days 1 and 19 and over 0-12 and 12-24 hour intervals after dosing on Day 11; a separate aliquot was taken from pooled 0-24 hour urine for urine creatinine concentration on Days 1, 11, and 19. Plasma and urine samples were analyzed using a validated LC-MS/MS method with a limit of quantification of 0.200 ng/mL and 1 ng/mL, respectively. The concentration of paliperidone in plasma and urine were calculated as the sum of the separate enantiomers. Based on the actual sampling times, the plasma and pharmacokinetic parameters were determined for paliperidone and its enantiomers.Safety evaluation was based on reports of adverse events, extrapyramidal symptoms (reported as adverse events or by Abnormal Involuntary Movement Scale [AIMS], Simpson Angus Scale [SAS], or Barnes Akathisia Rating Scale [BARS]), sedation (based on the Sedation Visual Analog Scale [VAS] and Sedation Questionnaire), and on change from baseline in clinical laboratory analyte values, vital sign measurements, orthostatic hypotension (based on the Orthostatic Hypotension Questionnaire), postural changes in blood pressure and heart rate, electrocardiograms, and physical examination findings. Paliperidone ER OROS tablet formulation (3 to 6 mg/day) to be taken orally. Patients were randomly assigned to receive either ER OROS paliperidone or placebo (4:1 ratio). All patients received a single dose of 3 mg ER OROS paliperidone (or placebo) on Day 1, a once daily regimen of 3 mg ER OROS paliperidone (or placebo) on Days 5 to 11, and a single dose of 6 mg ER OROS paliperidone (or placebo) on Day 19. All doses were administered in the fasted state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese and Caucasian patients. Japanese patients had to be born in Japan of Japanese parents and not to have lived outside of Japan for more than 5 years
* Normotensive (5 minute lying down systolic blood pressure of 100-139 mmHg and diastolic blood pressure of 60-89 mmHg)
* Body Mass Index of 18 to 25 kg/m2
* Considered healthy based on medical history, prestudy physical examination findings, electrocardiogram, and clinical laboratory evaluation of chemistry, hematology, and urinalysis values.

Exclusion Criteria:

* History of any significant cardiovascular, respiratory, neurologic, renal, hepatic, endocrine, psychiatric, or immunologic disorders
* Use of concomitant medication, except for paracetamol and hormonal contraceptives
* Has received an experimental drug and/or used an experimental medical device in the 60 days before the first dose.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2004-03; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of extended-release (ER) OROS paliperidone in healthy Japanese and Caucasian adults. Paliperidone plasma concentrations, time profiles and PK parameters after single and multiple dosing for Japanese and Caucasian patients.

SECONDARY OUTCOMES:
Pharmacogenomics: Relationships between composite genetic description or predicted observable traits and the pharmacokinetic parameters of paliperidone and its enantiomers were explored graphically.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Study evaluating and comparing single dose and multiple dose pharmacokinetics of ER OROS paliperidone in healthy Japanese and Caucasian adults — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=628&filename=CR004933_CSR.pdf